CLINICAL TRIAL: NCT01280175
Title: Pharmacokinetics and Lung Bioavailability of BDP/Formoterol HFA Fixed Combination After Single Administration in 12 Healthy Volunteers Using the Standard Actuator With or Without Charcoal Block or the Aerochamber Spacer.
Brief Title: Foster With or Without Charcoal Block or Aerochamber Plus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sara Collarini / Clinical Study Manager, Chiesi Farmaceutici
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FB/PS/14/163/06
Record Dates: First submitted 2011-01-17; First posted 2011-01-20 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
Keywords: BDP; Formoterol; pMDI; Aerochamber Plus; Charcoal
MeSH Terms: conditions — Anthrax | interventions — Metered Dose Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pMDI + charcoal block (Experimental): BDP/formoterol 100/6 µg pMDI with charcoal ingestion
  Interventions: Procedure: charcoal block
- pMDI + Aerochamber Plus (Experimental): BDP/formoterol 100/6 µg with Aerochamber Plus
  Interventions: Device: Aerochamber Plus spacer
- pMDI (Active Comparator): BDP/formoterol 100/g µg pMDI
  Interventions: Drug: pMDI standard actuator

INTERVENTIONS:
Procedure: charcoal block
  Arms: pMDI + charcoal block
Device: Aerochamber Plus spacer
  Arms: pMDI + Aerochamber Plus
Drug: pMDI standard actuator
  Arms: pMDI

SUMMARY:
The purpose of this study is to evaluate the systemic exposure of BDP, its metabolite beclomethasone 17-monopropionate (B17MP) and formoterol after inhalation of BDP/Formoterol 100/6 µg pMDI combination (CHF1535) using the standard actuator and charcoal block technique or using a Spacer (AeroChamber Plus, Trudell) in comparison with inhalation using the standard actuator

ELIGIBILITY:
Inclusion Criteria:

* Sex: male
* 18≤age≤45 years old
* BMI: 18≤BMI≤28 kg/m2
* Non-smokers
* Vital signs: SBP 100-139 mmHg, DBP 50-89, HR 50-90 bpm, measured after 5 min of rest in the sitting position
* Full comprehension: ability to use correctly the pMDI preparations; ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
* Informed Consent: signed written informed consent prior to inclusion in the study.

Exclusion Criteria:

* ECG (12 leads): clinically relevant abnormalities and/or QTc >450 msec;
* Physical findings: clinically relevant abnormal physical findings, which could interfere with the objectives of the study; in particular any abnormality in the lung functionality: FEV1 <80% predicted values according to European Respiratory Society basing upon Quanjer et al. (25)
* Laboratory analyses: clinically relevant abnormal laboratory values indicative of physical illness; in particular positive HIV1 and HIV2 serology and/or positive hepatitis serology indicating acute or chronic hepatitis B or C
* Allergy: ascertained or presumptive hypersensitivity to the active principles and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
* Diseases: relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases, that may interfere with the aim of the study
* Medications: medication, including OTC, during 2 weeks before the start of the study. Any known enzyme inducing drug or enzyme inhibitor must be stopped at least 2 months before study start
* Investigative drug trials: participation in the evaluation of any drug within 3 months prior to the screening
* Blood donation: blood donations during the 3 months prior to this study
* Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>2 drinks/day, defined according to USDA Dietary Guidelines 2005 (26)], caffeine (>5 cups coffee/tea/day) abuse or smoking
* Abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits within the past 4 weeks.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Systemic exposure and lung bioavailability of BDP, B17MP and formoterol. | from pre-dose until 12 h post-dose

SECONDARY OUTCOMES:
General tolerability and safety of the test product. | from pre-dose until 12 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rusca, MD, FMH, Principal Investigator — CROSS Research SA
Locations (1):
- CROSS Research SA, Arzo, Via F.A. Giorgioli, 14, Switzerland

REFERENCES:
- [Result] Singh D, Collarini S, Poli G, Acerbi D, Amadasi A, Rusca A. Effect of AeroChamber Plus on the lung and systemic bioavailability of beclometasone dipropionate/formoterol pMDI. Br J Clin Pharmacol. 2011 Dec;72(6):932-9. doi: 10.1111/j.1365-2125.2011.04024.x. PMID 21615456